CLINICAL TRIAL: NCT01217918
Title: APhase 1, Placebo-Controlled, Randomized, Parallel Group, Subject- And Investigator-Blind, Sponsor-Open Study To Assess The Safety, Tolerability, And Pharmacokinetics Of PH-797804 Following Multiple Escalating Oral Doses In Healthy Japanese Adult Subjects
Brief Title: Multiple Oral Doses Of PH-797804 In Healthy Japanese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A6631027
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: PH-797804; Japanese; Phase 1; multiple dose study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): PH-797804
  Interventions: Drug: 1 mg
- Cohort 2 (Experimental): PH-797804
  Interventions: Drug: 5 mg
- Cohotr 3 (Experimental): PH-797804
  Interventions: Drug: 10 mg

INTERVENTIONS:
Drug: 1 mg — 1 mg or placebo a material sparing tablet per day for 10 days
  Arms: Cohort 1
Drug: 5 mg — 5 mg or placebo as material sparing tablet per day for 10 days
  Arms: Cohort 2
Drug: 10 mg — 10 mg or placebo as a material sparing tablet per day for 10 days
  Arms: Cohotr 3

SUMMARY:
Study A6631027 will evaluate the safety, tolerability and pharmacokinetics of PH-797804 when administered to healthy Japanese subjects once a day (QD) for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Japanese

Exclusion Criteria:

* Subjects with clinically significant skin lesions
* Subjects with known tuberculosis infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events; of clinical findings on physical examination; and of clinical laboratory abnormalities. | Day 1 to Follow-up
Mean change from baseline in vital signs (blood pressure and heart rate) measurements | Baseline to Follow-up
Mean change from baseline in 12-lead ECG parameters | Baseline to Follow-up
Plasma PH-797804 Cmax, Cmin, Cavg(ss), Tmax, AUC(0-last), AUC(0-inf), AUC(0-tau), t1/2, CL/F, Vz/F, Rac, and Rac, Cmax | Days 1 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Culver City, California
  - Pfizer Investigational Site, Glendale, California

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631027&StudyName=Multiple%20Oral%20Doses%20Of%20PH-797804%20In%20Healthy%20Japanese%20Adult%20Subjects